CLINICAL TRIAL: NCT02241187
Title: Two Stage Study Of Single Dose PEGPH20 And Cetuximab In Patients With Pancreatic Adenocarcinoma Prior To Surgical Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cold Spring Harbor Laboratory (Other); Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-039
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: PEGPH20; Cetuximab; 14-039
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — PEGPH20; Cetuximab; Dynamic Contrast Enhanced Magnetic Resonance Imaging; Blood Specimen Collection

ARMS (1):
- PEGPH20 And Cetuximab (Experimental): 5 participants will undergo DW- & DCE-MRI for sequence parameter optimization. The 1st stage of the study, patients (n = 5) will have the option to undergo (DW-) & (DCE)-MRI for repeatability investigation & T1 mapping. Optional DW- & DCE-MRI will be repeated 2 to 5 days later, followed shortly by administration of 1 intravenous dose of cetuximab at 250 mg/m2/60 min. Pancreatic tumor resection will be performed 1 to 2 days later.Blood samples will be drawn at various time points. The resected tumor specimen will be studied. If deemed safe, we will proceed to the second stage of the study. Patients (n = 5) will have the option to undergo DW- & DCE-MRI. 1 to 3 days later, patients will receive 1 IV dose of PEGPH20 at 3 μg/kg/10 min. Optional DW- & DCE-MRI will be repeated 1 to 2 days after PEGPH20 administration, followed on that day by administration of 1 IV dose of cetuximab at 250 mg/m2/60 min. Pancreatic tumor resection will be performed 1 to 2 days later.
  Interventions: Drug: PEGPH20; Drug: Cetuximab; Device: DW & DCE-MRI; Other: blood draws

INTERVENTIONS:
Drug: PEGPH20
Drug: Cetuximab
Device: DW & DCE-MRI
Other: blood draws — Blood samples will be drawn at various time points.

SUMMARY:
This study has several purposes. DCE-MRI will be used to image the tumor. Safety of cetuximab given before surgery will be studied. Cetuximab delivery to the tumor will be studied. In Stage 2 of this study, the safety of cetuximab and PEGPH20 given before surgery will be studied. Also, the effects of PEGPH20 on tumors will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed PDAC. Pathologic confirmation is mandated before initiation of any protocol specified imaging studies or drug administrations. It is recognized that for some patients, histologic or cytologic confirmation of cancer may be obtained following study enrollment. Patient volunteers to the DW- and DCE-MRI sequence parameter optimization imaging portion of the study are eligible if they have any pancreatic lesion, histologic or cytologic confirmation of pathology is not required for this patient volunteer group.
* Radiographically resectable PDAC as adjudicated by MSKCC surgical oncologist without evidence of distant metastases by CT or by laparoscopy, if performed at the discretion of the surgeon.
* Age > 18 years.
* ECOG Performance Score of 0 - 2.
* Absolute neutrophil count > 1,500 cells/mm3
* Platelet count > 100,000 cells/mm3.
* Adequate renal function as evidenced by serum creatinine < 1.6 mg/dL.

  * INR < 1.5, unless patient is on therapeutic anticoagulation where a therapeutic INR is acceptable. Anticoagulation with low molecular weight heparin or warfarin, where medically indicated, is permitted.
* Patient volunteers for the DW- and DCE-MRI sequence parameter optimization portion of the study are exempt from criteria 2, 5, 6 and 8.
* Women of childbearing potential must have a negative pregnancy test prior to the administration of protocol specified interventions.
* Ability to understand informed consent and signing of written informed consent prior to initiation of protocol therapy.

Exclusion Criteria:

* Patients with histology other than adenocarcinoma, e.g., neuroendocrine cancer or acinar cancers, are ineligible.
* No prior therapy for pancreas cancer is allowed.
* Patients with metastatic or locally unresectable PDAC (resectability is as defined by MSKCC pancreatic surgeon and as outlined
* Active infection, with the exception of resolving cholangitis, will preclude enrollment on the study. Preoperative interventions can only be initiated when acute cholangitis has resolved.
* Patients with known hypersensitivity to any of the components of PEGPH20 or cetuximab.
* For patients who choose to undergo MRI imaging, hypersensitivity to MRI IV contrast media not suitable for pre-medication.
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication).
* Patients who have a history of venous or arterial thromboembolic events including pulmonary embolism, deep venous thrombosis and stroke.
* Patients who are pregnant or lactating
* For patients who choose to undergo MRI imaging patients who are ineligible for an MRI with contrast based on Radiology Department screening.
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or follow up procedures.
* Patient volunteers for the DW- and DCE-MRI sequence parameter optimization portion are exempt from criteria 12, 13, 14, 15, 16 and 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Yu, MD MSc, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 09/12/2014 Protocol Closed to Accrual N/A Primary Completion Date 09/13/2016 Recruitment Location is the medical clinic
Groups:
- PEGPH20 And Cetuximab: 5 participants will undergo DW- & DCE-MRI for sequence parameter optimization. The 1st stage of the study, patients (n = 5) will have the option to undergo (DW-) & (DCE)-MRI for repeatability investigation & T1 mapping. Optional DW- & DCE-MRI will be repeated 2 to 5 days later, followed shortly by administration of 1 intravenous dose of cetuximab at 250 mg/m2/60 min. Pancreatic tumor resection will be performed 1 to 2 days later.Blood samples will be drawn at various time points. The resected tumor specimen will be studied. If deemed safe, we will proceed to the second stage of the study. Patients (n = 5) will have the option to undergo DW- & DCE-MRI. 1 to 3 days later, patients will receive 1 IV dose of PEGPH20 at 3 μg/kg/10 min. Optional DW- & DCE-MRI will be repeated 1 to 2 days after PEGPH20 administration, followed on that day by administration of 1 IV dose of cetuximab at 250 mg/m2/60 min. Pancreatic tumor resection will be performed 1 to 2 days later.
  PEGPH20
  Cetuximab
Period: Overall Study
Arm/Group | PEGPH20 And Cetuximab
Started | 2
Completed | 0
Not Completed | 2
Not completed — Protocol closed due to lack of accrual. | 2

BASELINE CHARACTERISTICS:
Groups:
- PEGPH20 And Cetuximab: Participants have radiographically resectable Pancreatic ductal adenocarcinoma (PDAC) without evidence of distant metastases by CT or laparoscopy.
  However, the two participants accrued to this study were healthy participants.
Arm/Group | PEGPH20 And Cetuximab
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 64 [61 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Effects of PEGPH20
Description: administration on resectable pancreatic adenocarcinoma tumors. DW- and DCE-MRI and distribution of cetuximab will be used to study tumor permeability to small and larger molecules, respectively. Resected tumors will be carefully studied for evidence of stromal degradation.
Time Frame: 1 year
Population: The two participants accrued to this study were healthy participants. No participants were accrued on study for treatment. No data were collected.
Arm/Group | PEGPH20 And Cetuximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety of Administration of PEGPH20 and Cetuximab
Description: in close proximity to surgical resection of pancreatic adenocarcinoma. Safety with regards to operative and post-operative complications will be characterized.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | PEGPH20 And Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- PEGPH20 And Cetuximab: Participants have radiographically resectable Pancreatic ductal adenocarcinoma (PDAC) without evidence of distant metastases by CT or laparoscopy.
  All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were NOT monitored/assessed.
Arm/Group | PEGPH20 And Cetuximab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes